CLINICAL TRIAL: NCT02254681
Title: A Phase 2 Study of Low-Dose Fractionated Radiation Therapy to the Whole Liver in Combination With Gemcitabine and Cisplatin in Locally Advanced Mass-Forming Intrahepatic Cholangiocarcinoma
Brief Title: Low-Dose Radiation Therapy to the Whole Liver With Gemcitabine and Cisplatin in IHC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VPSR-1401
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: low-dose radiotherapy; gemcitabine; cisplatin; cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Gemcitabine; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Four three-week treatment cycles. Gemcitabine (1000 gm/m^2) and cisplatin (25 mg/m^2) administered on days one and eight of each cycle. Whole liver and portal lymph node basin low dose radiotherapy on days one, two, eight, and nine of each cycle.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Radiation: low dose radiotherapy

INTERVENTIONS:
Drug: Gemcitabine
  Other Names: Gemzar
Drug: Cisplatin
  Other Names: Platinol
Radiation: low dose radiotherapy — Whole liver and portal lymph node basin low dose radiotherapy

SUMMARY:
The overall goal of this study is to determine the safety and efficacy of combination treatment of low-dose fractionated radiation therapy with gemcitabine-cisplatin chemotherapy for locally advanced mass forming intra-hepatic cholangiocarcinoma.

DETAILED DESCRIPTION:
Intrahepatic cholangiocarcinoma (IHC) are cancers with pathologic features of biliary tract differentiation which arise from intrahepatic bile ducts and/or trans-differentiation of hepatocytes. IHC is the second most common primary liver cancer and its incidence and mortality rates are increasing both worldwide and in the United States. Approximately 80% of IHC in the Western hemisphere is the mass-forming type. Liver disease represents the major obstacle to long-term survival among patients with IHC. While partial hepatectomy offers the only hope of cure, less than 30% of IHC are resectable at initial presentation.2 Most patients have locally advanced disease (e.g. multi-focal tumors, major vascular invasion, local invasion of surrounding organs, and/or regional lymph node metastasis). Each of these factors portends poor 5-year survival (~20%) after surgical extirpation and are thus considered unresectable disease by most surgeons in the current era. Moreover, the liver is the most common site of disease recurrence after resection of IHC as 60-80% of initial disease recurrence occurs in the liver remnant.

Published response rates to preoperative or definitive radiation therapy (RT) for cholangiocarcinoma appear to be relatively high. For instance, a complete response proportion of 48% was recently reported for perihilar cholangiocarcinoma patients who received preoperative chemoradiation followed by liver transplant. Moreover, small series have demonstrated superior progression free and overall survival with the combination of external beam RT and chemotherapy compared to that derived from chemotherapy alone for many unresectable hepatic malignancies, including IHC, colorectal cancer liver metastases, and hepatocellular carcinoma. For example, addition of external beam RT to cisplatin chemotherapy was associated with prolonged progression free (median 4.3 vs. 1.9 months, p=0.001) and overall (median 9.3 vs. 6.2 months, p=0.048) survival compared to cisplatin alone among 92 total patients with unresectable IHC. Traditional thoughts in radiation biology of tumors suggested that doses of at least 1.2 Gy were required to overcome the initial shoulder of the cell survival curve. In practice, the standard dose per fraction is considered to be 0.015-0.022 Gy per fraction although the vast majority of patients are treated with either 1.8 Gy or 2 Gy fractions.

Laboratory and clinical data suggest that a new paradigm using LDFRT as a chemopotentiator may allow full-dose drug therapy with improved efficacy without adding to the toxicity of the systemic treatment. This chemopotentiating effect is possible through a phenomenon known as hyper-radiation sensitivity (HRS) by which there is more effective tumor cell killing than would be predicted when using doses per fraction below 1 Gy. This is followed by a change in slope of the survival response with increasing doses per fraction, indicating increased radioresistance (IRR). This HRS phenomenon was first described by Joiner and colleagues in the Gray Laboratory in 1986 and has since been well described by a number of other laboratories. It also has been documented in the clinical setting; in a study by Harney et al., patients with paired cutaneous metastases from sarcoma and melanoma had longer time to tumor regrowth after LDFRT than with conventional radiation. In vitro studies have established a link between HRS/IRR and evasion of the early G2/M cell cycle checkpoint. Exaggerated HRS/IRR responses were found for enriched populations of G2 phase cells in one study, indicating that the mechanism likely involved events in the G2 phase of the cell cycle. Two G2 checkpoints have been described, and the more recently discovered "early" checkpoint is rapidly activated after radiation exposure. It is believed to prevent cell cycle progression through G2 of cells with unrepaired radiation-induced DNA damage. The signaling cascade regulating the early G2/M checkpoint is initiated through ATM activity. Joiner and colleagues have shown that inhibition of ChK1 and Chk2, two proteins integral to the G2/M transition, can influence the cell-cycle response to low-dose radiation. It is believed that failure of the cell to repair DNA damage in G2-phase cells leads to increased apoptosis. Nonetheless, inhibition of ChK1 and ChK2 also lead to IRR at radiation doses > 0.2 Gy. This is consistent with reports indicating that low dose radiation can stimulate repair of DNA damage. Interestingly, low dose radiation can also stimulate antioxidant capacity, apoptosis, and induction of immune responses, which collectively may provide effective local tumor control. In addition, hypoxia and nitric oxide levels can also affect cells sensitivity to radiation. Reduction of nitric oxide level enhances the radiosensitivity of hypoxic non-small cell lung cancer. Therefore, the identification of cellular pathways that are responsive to low dose radiation and their contribution to chemopotentiation is highly significant because this will provide a better measurement of the therapeutic response and contribute to the rational design of mechanism-based clinical trials.

Based on promising preclinical data, clinical studies have been performed in a variety of cancer types with LDFRT in addition to standard chemotherapy. Investigators at the University of Kentucky published their experience using carboplatin and paclitaxel with 4 fractions of 0.8 Gy each in locally advanced head and neck cancer patients. They observed toxicities similar to those expected from chemotherapy alone and concluded that the addition of LDFRT was "extremely well tolerated." Moreover, they reported excellent response rates. Regine et al. conducted a phase I trial of low dose abdominal RT (0.6 vs. 0.7 Gy fractions, total 8 fractions) and gemcitabine 1,250 mg/m2 among patients with unresectable pancreatic/small bowel carcinomas. The authors concluded that abdominal LDFRT using 0.6 Gy fractions was well tolerated when given concurrently with full-dose gemcitabine. A multi-institutional phase II trial using this regimen suggested improved efficacy of the combined regimen in improving overall survival. Sixty-one percent of enrolled patients experienced at least stable disease, and median survival in this poor prognosis population was 13 months. More importantly, no additional toxicity was observed with LDFRT other than that expected from the high dose of gemcitabine (personal communication, manuscript in preparation). More recently, Wrenn et al. demonstrated tolerability of concomitant low-dose whole-abdominal RT and full-dose cisplatin in optimally debulked stage III/IV endometrial cancer patients.

Currently, there are no prospective studies evaluating the efficacy of concomitant gem-cis and RT for locally advanced IHC regarding disease response or post-operative intrahepatic disease recurrence. Prior full dose external beam RT is an accepted contraindication to liver resection due to development of advanced fibrosis and intrahepatic biliary sclerosis. However, no studies have evaluated the influence of preoperative LDFRT on outcomes after partial hepatectomy. Case reports of safe liver resection after antecedent radioembolization suggest that LDFRT may not adversely affect postoperative outcomes. LDFRT to the entire liver and portal lymph node basin is advantageous compared to tumor directed therapy as the former treats occult disease representing the most common site of disease recurrence after partial hepatectomy and progression after chemotherapy.

Based on data from the ABC trial establishing gem-cis as the standard of care for locally advanced and/or metastatic cholangiocarcinoma, the primary goal of this phase II study is to explore the safety and efficacy of using a combination of LDFRT as a chemopotentiator and concurrent gem-cis for mass-forming IHC.

The pivotal Advanced Biliary Tract Cancer (ABC) Trial established combination gemcitabine-cisplatin (gem-cis) therapy as the standard of care for patients with locally advanced and/or metastatic IHC. While the majority of patients experience initial disease stabilization after therapy (e.g. stable disease, partial response, or complete response) partial or complete response occurs in only approximately 20% of patients. Smaller trials comprising other chemotherapeutics with or without anti-biologic agents report similar results. Moreover, disease stabilization is short lived with median progression free survival of only six-eight months. Thus, there is a pressing need for more effective liver directed therapy for locally advanced disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of mass-forming IHC. OR
* Histologic diagnosis of adenocarcinoma of the liver in setting of negative colonoscopy, upper endoscopy, mammography (females), or cross-sectional imaging for primary disease.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as ≥10 mm (≥1 cm) with spiral CT scan, MRI. See Section 8 for the evaluation of measurable disease.
* Locally advanced disease (portal lymph node disease, multifocal intrahepatic lesions, or major vascular invasion) AND no evidence of omental, peritoneal, or pelvic metastases.
* Other sites of metastatic disease (e.g. lung, distant lymph nodes, bone) are allowed.
* No prior chemotherapy, radiotherapy, or surgical therapy.
* ECOG performance status ≤ 1 (Karnofsky ≥70%). See Appendix A.
* Life expectancy of greater than six months.
* Patients must have normal organ and marrow function as defined below:
* leukocytes≥3,000/mcL
* absolute neutrophil count≥1,500/mcL
* platelets ≥100,000/mcL
* hemoglobin≥9.0 g/dL
* total bilirubin≤2.0 mg/dL
* AST(SGOT)/ALT(SGPT)≤3 × institutional upper limit of normal
* creatinine within normal institutional limits OR
* creatinine clearance≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* int'l normalized ratio<1.8
* systolic blood pressure≤160 mmHg
* diastolic blood pressure ≥90 mmHg
* For women of child-bearing potential, negative serum pregnancy test within 14 days prior to registration.
* Women of childbearing age and male participants.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior chemotherapy, surgical therapy, or radiotherapy for IHC.
* Patients who are receiving any other investigational agents or have been treated with any other therapeutic clinical protocols within 30 days prior to study entry or during participation in the study.
* Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine or cisplatin.
* Prior invasive malignancy (except for non-melanomatous skin cancer, low grade prostate cancer, and in situ cervical cancer) unless disease free for ≥ two years.
* Periductal infiltrating, intraductal, or poorly differentiated neuroendocrine (e.g. high grade, small, or large cell) tumor histology.
* Prior abdominal radiotherapy.
* Cirrhosis, primary sclerosing cholangitis, hepatitis viral infection (documented by positive serology and antigen serologic testing), or other background liver diseases.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection; unstable angina and/or congestive heart failure within the last 6 months; transmural myocardial infarction within the last 6 months; New York Heart Association grade II or greater congestive heart failure requiring hospitalization within 12 months prior to registration; history of stroke, cerebral vascular accident or transient ischemic attack within 6 months; serious and inadequately controlled cardiac arrhythmia; significant vascular disease (e.g.;, high risk aortic aneurysm, history of aortic dissection) or clinically significant peripheral vascular disease; evidence of bleeding diathesis or coagulopathy; serious or non-healing wound, ulcer, or bone fracture or history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess, major surgical procedure or significant traumatic injury within 28 days prior to registration; bacterial or fungal infection requiring intravenous antibiotics at the time of registration; chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration; active connective tissue disorders, such as lupus or scleroderma, that in the opinion of the treating physician may put the patient at high risk for radiation toxicity; any other major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy; cognitive impairment that precludes a patient from acting as his or her own agent to provide informed consent.
* Pregnant or breast feeding women.
* Men and women of childbearing potential who are sexually active and not willing/able to use medically acceptable forms of contraception.
* Acquired immune deficiency syndrome (AIDS) based upon current CDC definition. Note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol are significantly immunosuppressive.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinevas K Reddy, MD, Principal Investigator — Allina Health System
Locations (1):
- Virginia Piper Cancer Institute, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Bridgewater J, Galle PR, Khan SA, Llovet JM, Park JW, Patel T, Pawlik TM, Gores GJ. Guidelines for the diagnosis and management of intrahepatic cholangiocarcinoma. J Hepatol. 2014 Jun;60(6):1268-89. doi: 10.1016/j.jhep.2014.01.021. Epub 2014 Mar 27. No abstract available. PMID 24681130
- [Background] Ilyas SI, Gores GJ. Pathogenesis, diagnosis, and management of cholangiocarcinoma. Gastroenterology. 2013 Dec;145(6):1215-29. doi: 10.1053/j.gastro.2013.10.013. Epub 2013 Oct 15. PMID 24140396
- [Background] de Jong MC, Nathan H, Sotiropoulos GC, Paul A, Alexandrescu S, Marques H, Pulitano C, Barroso E, Clary BM, Aldrighetti L, Ferrone CR, Zhu AX, Bauer TW, Walters DM, Gamblin TC, Nguyen KT, Turley R, Popescu I, Hubert C, Meyer S, Schulick RD, Choti MA, Gigot JF, Mentha G, Pawlik TM. Intrahepatic cholangiocarcinoma: an international multi-institutional analysis of prognostic factors and lymph node assessment. J Clin Oncol. 2011 Aug 10;29(23):3140-5. doi: 10.1200/JCO.2011.35.6519. Epub 2011 Jul 5. PMID 21730269
- [Background] Endo I, Gonen M, Yopp AC, Dalal KM, Zhou Q, Klimstra D, D'Angelica M, DeMatteo RP, Fong Y, Schwartz L, Kemeny N, O'Reilly E, Abou-Alfa GK, Shimada H, Blumgart LH, Jarnagin WR. Intrahepatic cholangiocarcinoma: rising frequency, improved survival, and determinants of outcome after resection. Ann Surg. 2008 Jul;248(1):84-96. doi: 10.1097/SLA.0b013e318176c4d3. PMID 18580211
- [Background] Lang H, Sotiropoulos GC, Sgourakis G, Schmitz KJ, Paul A, Hilgard P, Zopf T, Trarbach T, Malago M, Baba HA, Broelsch CE. Operations for intrahepatic cholangiocarcinoma: single-institution experience of 158 patients. J Am Coll Surg. 2009 Feb;208(2):218-28. doi: 10.1016/j.jamcollsurg.2008.10.017. PMID 19228533
- [Background] Choi SB, Kim KS, Choi JY, Park SW, Choi JS, Lee WJ, Chung JB. The prognosis and survival outcome of intrahepatic cholangiocarcinoma following surgical resection: association of lymph node metastasis and lymph node dissection with survival. Ann Surg Oncol. 2009 Nov;16(11):3048-56. doi: 10.1245/s10434-009-0631-1. Epub 2009 Jul 22. PMID 19626372
- [Background] Paik KY, Jung JC, Heo JS, Choi SH, Choi DW, Kim YI. What prognostic factors are important for resected intrahepatic cholangiocarcinoma? J Gastroenterol Hepatol. 2008 May;23(5):766-70. doi: 10.1111/j.1440-1746.2007.05040.x. Epub 2007 Sep 12. PMID 17868336
- [Background] Nakagohri T, Kinoshita T, Konishi M, Takahashi S, Gotohda N. Surgical outcome and prognostic factors in intrahepatic cholangiocarcinoma. World J Surg. 2008 Dec;32(12):2675-80. doi: 10.1007/s00268-008-9778-3. PMID 18843437
- [Background] Tamandl D, Herberger B, Gruenberger B, Puhalla H, Klinger M, Gruenberger T. Influence of hepatic resection margin on recurrence and survival in intrahepatic cholangiocarcinoma. Ann Surg Oncol. 2008 Oct;15(10):2787-94. doi: 10.1245/s10434-008-0081-1. Epub 2008 Aug 7. PMID 18685896
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Background] Woo SM, Lee WJ, Kim JH, Kim DH, Han SS, Park SJ, Kim TH, Lee JH, Koh YH, Hong EK. Gemcitabine plus cisplatin versus capecitabine plus cisplatin as first-line chemotherapy for advanced biliary tract cancer: a retrospective cohort study. Chemotherapy. 2013;59(3):232-8. doi: 10.1159/000354539. Epub 2013 Dec 13. PMID 24356333
- [Background] Alberts SR, Al-Khatib H, Mahoney MR, Burgart L, Cera PJ, Flynn PJ, Finch TR, Levitt R, Windschitl HE, Knost JA, Tschetter LK. Gemcitabine, 5-fluorouracil, and leucovorin in advanced biliary tract and gallbladder carcinoma: a North Central Cancer Treatment Group phase II trial. Cancer. 2005 Jan 1;103(1):111-8. doi: 10.1002/cncr.20753. PMID 15558814
- [Background] Jensen LH, Lindebjerg J, Ploen J, Hansen TF, Jakobsen A. Phase II marker-driven trial of panitumumab and chemotherapy in KRAS wild-type biliary tract cancer. Ann Oncol. 2012 Sep;23(9):2341-2346. doi: 10.1093/annonc/mds008. Epub 2012 Feb 23. PMID 22367707
- [Background] Lubner SJ, Mahoney MR, Kolesar JL, Loconte NK, Kim GP, Pitot HC, Philip PA, Picus J, Yong WP, Horvath L, Van Hazel G, Erlichman CE, Holen KD. Report of a multicenter phase II trial testing a combination of biweekly bevacizumab and daily erlotinib in patients with unresectable biliary cancer: a phase II Consortium study. J Clin Oncol. 2010 Jul 20;28(21):3491-7. doi: 10.1200/JCO.2010.28.4075. Epub 2010 Jun 7. PMID 20530271
- [Background] Darwish Murad S, Kim WR, Harnois DM, Douglas DD, Burton J, Kulik LM, Botha JF, Mezrich JD, Chapman WC, Schwartz JJ, Hong JC, Emond JC, Jeon H, Rosen CB, Gores GJ, Heimbach JK. Efficacy of neoadjuvant chemoradiation, followed by liver transplantation, for perihilar cholangiocarcinoma at 12 US centers. Gastroenterology. 2012 Jul;143(1):88-98.e3; quiz e14. doi: 10.1053/j.gastro.2012.04.008. Epub 2012 Apr 12. PMID 22504095
- [Background] Kim YI, Park JW, Kim BH, Woo SM, Kim TH, Koh YH, Lee WJ, Kim CM. Outcomes of concurrent chemoradiotherapy versus chemotherapy alone for advanced-stage unresectable intrahepatic cholangiocarcinoma. Radiat Oncol. 2013 Dec 21;8:292. doi: 10.1186/1748-717X-8-292. PMID 24359879
- [Background] Ben-Josef E, Normolle D, Ensminger WD, Walker S, Tatro D, Ten Haken RK, Knol J, Dawson LA, Pan C, Lawrence TS. Phase II trial of high-dose conformal radiation therapy with concurrent hepatic artery floxuridine for unresectable intrahepatic malignancies. J Clin Oncol. 2005 Dec 1;23(34):8739-47. doi: 10.1200/JCO.2005.01.5354. PMID 16314634
- [Background] Servajean C, Gilabert M, Piana G, Monges G, Delpero JR, Brenot I, Raoul JL. One case of intrahepatic cholangiocarcinoma amenable to resection after radioembolization. World J Gastroenterol. 2014 May 7;20(17):5131-4. doi: 10.3748/wjg.v20.i17.5131. PMID 24803830
- [Background] Vouche M, Lewandowski RJ, Atassi R, Memon K, Gates VL, Ryu RK, Gaba RC, Mulcahy MF, Baker T, Sato K, Hickey R, Ganger D, Riaz A, Fryer J, Caicedo JC, Abecassis M, Kulik L, Salem R. Radiation lobectomy: time-dependent analysis of future liver remnant volume in unresectable liver cancer as a bridge to resection. J Hepatol. 2013 Nov;59(5):1029-36. doi: 10.1016/j.jhep.2013.06.015. Epub 2013 Jun 25. PMID 23811303
- [Background] Inarrairaegui M, Pardo F, Bilbao JI, Rotellar F, Benito A, D'Avola D, Herrero JI, Rodriguez M, Marti P, Zozaya G, Dominguez I, Quiroga J, Sangro B. Response to radioembolization with yttrium-90 resin microspheres may allow surgical treatment with curative intent and prolonged survival in previously unresectable hepatocellular carcinoma. Eur J Surg Oncol. 2012 Jul;38(7):594-601. doi: 10.1016/j.ejso.2012.02.189. Epub 2012 Mar 21. PMID 22440743
- [Background] Mullen JT, Ribero D, Reddy SK, Donadon M, Zorzi D, Gautam S, Abdalla EK, Curley SA, Capussotti L, Clary BM, Vauthey JN. Hepatic insufficiency and mortality in 1,059 noncirrhotic patients undergoing major hepatectomy. J Am Coll Surg. 2007 May;204(5):854-62; discussion 862-4. doi: 10.1016/j.jamcollsurg.2006.12.032. Epub 2007 Feb 15. PMID 17481498
- [Background] Marples B, Wouters BG, Collis SJ, Chalmers AJ, Joiner MC. Low-dose hyper-radiosensitivity: a consequence of ineffective cell cycle arrest of radiation-damaged G2-phase cells. Radiat Res. 2004 Mar;161(3):247-55. doi: 10.1667/rr3130. PMID 14982490
- [Background] Short SC, Woodcock M, Marples B, Joiner MC. Effects of cell cycle phase on low-dose hyper-radiosensitivity. Int J Radiat Biol. 2003 Feb;79(2):99-105. PMID 12569013
- [Background] Joiner MC, Marples B, Lambin P, Short SC, Turesson I. Low-dose hypersensitivity: current status and possible mechanisms. Int J Radiat Oncol Biol Phys. 2001 Feb 1;49(2):379-89. doi: 10.1016/s0360-3016(00)01471-1. PMID 11173131
- [Background] Kunos CA, Sill MW, Buekers TE, Walker JL, Schilder JM, Yamada SD, Waggoner SE, Mohiuddin M, Fracasso PM. Low-dose abdominal radiation as a docetaxel chemosensitizer for recurrent epithelial ovarian cancer: a phase I study of the Gynecologic Oncology Group. Gynecol Oncol. 2011 Feb;120(2):224-8. doi: 10.1016/j.ygyno.2010.10.018. PMID 21075438
- [Background] Arnold SM, Regine WF, Ahmed MM, Valentino J, Spring P, Kudrimoti M, Kenady D, Desimone P, Mohiuddin M. Low-dose fractionated radiation as a chemopotentiator of neoadjuvant paclitaxel and carboplatin for locally advanced squamous cell carcinoma of the head and neck: results of a new treatment paradigm. Int J Radiat Oncol Biol Phys. 2004 Apr 1;58(5):1411-7. doi: 10.1016/j.ijrobp.2003.09.019. PMID 15050317
- [Background] Harney J, Short SC, Shah N, Joiner M, Saunders MI. Low dose hyper-radiosensitivity in metastatic tumors. Int J Radiat Oncol Biol Phys. 2004 Jul 15;59(4):1190-5. doi: 10.1016/j.ijrobp.2003.12.029. PMID 15234055
- [Background] Joiner MC, Denekamp J. The effect of small radiation doses on mouse skin. Br J Cancer Suppl. 1986;7:63-6. No abstract available. PMID 3459542
- [Background] Krueger SA, Wilson GD, Piasentin E, Joiner MC, Marples B. The effects of G2-phase enrichment and checkpoint abrogation on low-dose hyper-radiosensitivity. Int J Radiat Oncol Biol Phys. 2010 Aug 1;77(5):1509-17. doi: 10.1016/j.ijrobp.2010.01.028. PMID 20637979
- [Background] Marples B, Wouters BG, Joiner MC. An association between the radiation-induced arrest of G2-phase cells and low-dose hyper-radiosensitivity: a plausible underlying mechanism? Radiat Res. 2003 Jul;160(1):38-45. doi: 10.1667/rr3013. PMID 12816521
- [Background] Regine WF, Hanna N, Garofalo MC, Doyle A, Arnold S, Kataria R, Sims J, Tan M, Mohiuddin M. Low-dose radiotherapy as a chemopotentiator of gemcitabine in tumors of the pancreas or small bowel: a phase I study exploring a new treatment paradigm. Int J Radiat Oncol Biol Phys. 2007 May 1;68(1):172-7. doi: 10.1016/j.ijrobp.2006.11.045. Epub 2007 Feb 2. PMID 17276612
- [Background] Wrenn DC, Saigal K, Lucci JA 3rd, Pearson MJ, Simpkins F, Schuman S, Twiggs LB, Walker GR, Wolfson AH. A Phase I Study using low-dose fractionated whole abdominal radiotherapy as a chemopotentiator to full-dose cisplatin for optimally debulked stage III/IV carcinoma of the endometrium. Gynecol Oncol. 2011 Jul;122(1):59-62. doi: 10.1016/j.ygyno.2011.03.007. Epub 2011 Apr 6. PMID 21474169
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 subjects recruited from 9/2014-12/2015
Groups:
- Treatment: Four three-week treatment cycles. Gemcitabine (1000 gm/m^2) and cisplatin (25 mg/m^2) administered on days one and eight of each cycle. Whole liver and portal lymph node basin low dose radiotherapy on days one, two, eight, and nine of each cycle.
  Gemcitabine
  Cisplatin
  Low dose whole liver and portal lymph node basin radiotherapy
Period: Overall Study
Arm/Group | Treatment
Started | 6
Completed | 0
Not Completed | 6
Not completed — Lack of Efficacy | 6

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Radiographic Disease Response After Combination Low-dose Radiotherapy and Gemcitabine-cisplatin.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD), At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: 16 weeks after treatment start
Population: decision was made to close the study due to the futility of the regimen in the first 6 subjects, as well as the lack of funding to complete the study.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment: Four three-week treatment cycles. Gemcitabine (1000 gm/m^2) and cisplatin (25 mg/m^2) administered on days one and eight of each cycle. Whole liver and portal lymph node basin low dose radiotherapy on days one, two, eight, and nine of each cycle.
  Gemcitabine
  Cisplatin
  Low dose whole liver and portal lymph node basin radiotherapy
  decision was made to close the study due to the futility of the regimen in the first 6 subjects, as well as the lack of funding to complete the study.
Arm/Group | Treatment
Number analyzed (Participants) | 6
Participants
  Stable Disease | 5
  Partial Response | 1

2. Primary Outcome: Number of Participants With Adverse Events.
Description: Number of participants with adverse events during combined low-dose radiotherapy and gemcitabine-cisplatin treatment.
Time Frame: up to 16 weeks after treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 6
Participants
  Study related Adverse events | 6
  No study related Adverse Events | 0

3. Secondary Outcome: Number of Participants With Post-operative Complications After Partial Hepatectomy After Antecedent Combination Low-dose Radiotherapy and Gemcitabine-cisplatin.
Description: Measured post-operative complications include (but not limited to) bile leak, liver failure, ascites, infection, any organ failure or insufficiency, venous thromboembolism, and mortality.
Time Frame: up to 90 days after partial hepatectomy
Population: 1 of 6 subjects had surgery therefore only 1 subject was analyzed for post-operative complications.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 1
Participants | 1

4. Secondary Outcome: Number of Participants With Histologic Disease Response After Combination Low-dose Radiotherapy and Gemcitabine-cisplatin.
Description: Tumor tissue will be obtained by either biopsy or liver resection after combination chemoradiotherapy. Histologic response will be determined by extent of viable tumor, tumor necrosis, and surrounding fibrosis.
Time Frame: 16 weeks after start of first treatment
Population: data not collected
Arm/Group | Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Injury to the Background Liver After Combination Low-dose Radiotherapy and Gemcitabine-cisplatin.
Description: Background (non-tumor bearing) liver tissue will be obtained by either biopsy or liver resection after combination chemoradiotherapy. Histologic markers of Radiation Induced Liver disease will be measured.
Time Frame: 16 weeks after start of first treatment.
Population: data not collected
Arm/Group | Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With Intrahepatic Recurrence After Partial Hepatectomy With Antecedent Combination Low-dose Radiotherapy and Gemcitabine-cisplatin.
Description: To determine the number of participants with Intrahepatic recurrence assessed by RECIST criteria using MRI of the abdomen with intravenous gadolinium contrast.
Time Frame: From date of partial hepatectomy until date of first documented recurrence or date of death from any cause, assessed up to 24 months.
Population: Only 1 of the 6 subjects had surgery to assess recurrence after hepatectomy.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment: Four three-week treatment cycles. Gemcitabine (1000 gm/m^2) and cisplatin (25 mg/m^2) administered on days one and eight of each cycle. Whole liver and portal lymph node basin low dose radiotherapy on days one, two, eight, and nine of each cycle.
  Gemcitabine
  Cisplatin
  liver and portal lymph node low dose Radiotherapy
Arm/Group | Treatment
Number analyzed (Participants) | 1
Participants | 1

7. Secondary Outcome: Number of Participants With Intrahepatic Disease Progression After Treatment With Combination Low-dose Radiotherapy and Gemcitabine-cisplatin.
Description: To determine the number of participants with Intrahepatic disease progression assessed by MRI of the abdomen with intravenous gadolinium contrast using RECIST criteria.
Time Frame: From date of first treatment until date of first documented progression or date of death from any cause, which ever comes first, assessed up to 24 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: 1.5 years
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 3/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=6)
cholelithiasis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=6)
anemia (Blood and lymphatic system disorders) | 1 (1)
neutropenia (Investigations) | 4 (4)
thrombocytopenia (Investigations) | 2 (2)
hypomagnesemia (Metabolism and nutrition disorders) | 3 (5)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2)
pain (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes